CLINICAL TRIAL: NCT07388836
Title: A Multicenter, Randomized, Phase II Clinical Trial to Optimize the Timing of Immune Checkpoint Inhibitor Administration During Neoadjuvant Chemotherapy in Patients With Locally Advanced Nasopharyngeal Carcinoma
Brief Title: Timing Optimization of Immunotherapy During Neoadjuvant Chemotherapy for Locally Advanced Nasopharyngeal Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Huang Chaobin, Professor, Fujian Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2026-01-15
Record Dates: First submitted 2026-01-15; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Locally Advanced Nasopharyngeal Carcinoma
MeSH Terms: interventions — toripalimab

STUDY DESIGN:
Intervention Model Description: Participants will be assigned in a 1:1:1 ratio to three parallel arms receiving gemcitabine and cisplatin chemotherapy combined with toripalimab administered on Day 1 (control), Day 5 (exploratory), or Day 9 (experimental).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Arm (No Intervention): Participants receive gemcitabine and cisplatin chemotherapy combined with toripalimab administered on Day 1 of each 21-day cycle for 3 cycles.
- Experimental Arm (Experimental): Participants receive gemcitabine and cisplatin chemotherapy combined with toripalimab administered on Day 9 of each 21-day cycle for 3 cycles.
  Interventions: Drug: Toripalimab
- Exploratory Arm (Experimental): Participants receive gemcitabine and cisplatin chemotherapy combined with toripalimab administered on Day 5 of each 21-day cycle for 3 cycles. This arm is exploratory in nature with a smaller sample size.
  Interventions: Drug: Toripalimab

INTERVENTIONS:
Drug: Toripalimab — Toripalimab 240 mg IV on Day 9, every 21-day cycle, for 3 cycles.
  Arms: Experimental Arm
Drug: Toripalimab — Toripalimab 240 mg IV on Day 5 depending, every 21-day cycle, for 3 cycles.
  Arms: Exploratory Arm

SUMMARY:
This is a multicenter, open-label, randomized phase II clinical trial designed to evaluate the optimal timing of toripalimab administration during neoadjuvant chemotherapy in patients with locoregionally advanced nasopharyngeal carcinoma. Participants will receive gemcitabine and cisplatin (GP) chemotherapy combined with toripalimab administered on different days (Day 1, Day 5, or Day 9) to compare treatment responses. The neoadjuvant phase includes 3 cycles of 21 days each, followed by concurrent chemoradiotherapy. The estimated enrollment period is from March 2026 to March 2028.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years

Histologically confirmed locoregionally advanced nasopharyngeal carcinoma (AJCC/UICC 8th edition stage II-III)

At least one measurable target lesion per RECIST 1.1

ECOG performance status of 0-1

Estimated life expectancy ≥ 6 months

Adequate hematologic, hepatic, renal, and coagulation function

Negative pregnancy test for women of childbearing potential

Willingness to use effective contraception during the study and for 12 months after treatment

Signed informed consent

Willing and able to comply with study procedures

Not participating in any other interventional clinical trials during the study period

Exclusion Criteria:

* re first dose

Active or suspected autoimmune disease requiring systemic treatment

Ongoing systemic immunosuppressive therapy

Active hepatitis B, hepatitis C, HIV infection, or other serious infections

History of another malignancy within 5 years (except non-melanoma skin cancer or in situ cervical cancer)

Pregnant or breastfeeding women

Inability or unwillingness to use contraception as required

Life expectancy < 6 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Complete Response Rate | After 2 cycles of neoadjuvant therapy (21-28 days for each cycle)
  The proportion of participants achieving complete response (CR) after 2 cycles of neoadjuvant chemotherapy combined with toripalimab, as assessed by RECIST or institutional imaging criteria.

SECONDARY OUTCOMES:
Objective Response Rate | After 2 cycles of neoadjuvant therapy (21-28 days for each cycle)
  The proportion of participants achieving complete response (CR) or partial response (PR) after 2 cycles of neoadjuvant chemo-immunotherapy.
Disease Control Rate | After 2 cycles of neoadjuvant therapy (21-28 days for each cycle)
  The proportion of participants with CR, PR, or stable disease (SD) after 2 cycles of neoadjuvant chemo-immunotherapy.
EBV DNA Clearance Rate | After 2 cycles of neoadjuvant therapy (21-28 days for each cycle)
  The proportion of participants with undetectable plasma Epstein-Barr virus (EBV) DNA levels after 2 cycles of neoadjuvant chemo-immunotherapy.
Incidence of Grade ≥3 Treatment-Related Adverse Events | From first dose until 30 days after the end of neoadjuvant therapy
  The frequency of treatment-related adverse events (AEs) of grade 3 or higher, according to CTCAE version 5.0.

IPD SHARING:
Plan to Share IPD: No